CLINICAL TRIAL: NCT06624007
Title: Application of Pediatric Nursing Excellence Model on Nurses, Performance Regarding Care of Children Undergoing Orthopedic Surgeries
Brief Title: Applying Pediatric Nursing Excellence Model to Nurses in Orthopedic Surgery Care of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Nadia Elsharkawy, Associate Professor- Department of Maternal and Newborn Health Nursing - College of Nursing- Jouf University, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 358-12-2023
Record Dates: First submitted 2024-09-21; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pediatric ALL; Nurse's Role; Surgery
Keywords: Pediatric; Nursing Excellence Model; Nurses Performance
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Models, Biological

STUDY DESIGN:
Intervention Model Description: Group A: intervention group: Nurses who will apply Pediatric nursing excellence(PNE) model for children having orthopedic surgery.
  Group B: Control group: Nurses who will provide routine care only for children having orthopedic surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will interview participants, explain the purpose of the study and they will ask them to sign the consent. intervention group will apply Pediatric nursing excellence(PNE) model for children having orthopedic surgery, while the control group will provide routine care only for children having orthopedic surgery.
  They will randomly assign in two intervention and control groups (50 each) using a computer-generated table of random numbers and they are unaware of which group they have been assigned to as well as the outcome assessor is unaware
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A (Experimental): They will apply pediatric Nursing Excellence (PNE) model for children having orthopedic surgery
  Interventions: Other: pediatric Nursing Excellence (PNE) model
- Control group (No Intervention): They will provide routine care for children having orthopedic surgery

INTERVENTIONS:
Other: pediatric Nursing Excellence (PNE) model — The intervention group will apply pediatric Nursing Excellence (PNE) model included 28 Likert-type questions to assess nurses' general excellence level regarding the care of children undergoing orthopedic surgeries grouped under five main categories including engagement, values, principles, care delivery and continuous improvement.
  Arms: Intervention A

SUMMARY:
Problem description: Orthopedic surgeries are common in pediatric orthopedics, treating various conditions resulting from developmental, genetic, neoplastic, nutritional, infection, neurological, or physical injuries. The Pediatric Nursing Excellence model helps nurses provide optimal care, improve childcare systems, and deliver high-quality care. It also helps nurses identify trends in specialty nursing excellence. The study aims to evaluate the application of the Pediatric Nursing Excellence Model on nurses' performance regarding the care of children undergoing orthopedic surgeries. Methodology: Randomized Controlled Trial will be conducted using a sample of 100 nurses working in the pediatric inpatient surgical unit of Tanta University Hospital. Three tools will be used for data collection: a knowledge assessment questionnaire, an orthopedic surgeries nurse practice observational checklist, and the Pediatric Nursing Excellence (PNE) model. All study participants will randomly assign to two intervention and control groups (50 each) using a computer-generated table of random numbers. Pediatric Nursing Excellence Model will be applied for the intervention group. The Control group receive routine care. The study participants will be informed about the nature and aim of the study with assuring confidentiality and anonymity. Expected outcome: Nurses who will participate in the pediatric nursing excellence (PNE) model application are expected to have an improvement in their performance regarding care of children undergoing orthopedic surgeries.

DETAILED DESCRIPTION:
Orthopedic surgeries are more prevalent among children and are the most conclusive approach of treatment in pediatric orthopedics addressing wide range of conditions and deformities resulting from developmental or genetic disorders, neoplastic disorders, nutritional disorders, infection, neurological conditions, or physical injuries that necessitate extensive surgical intrusions to recover musculoskeletal alignment, functional abilities, control pain, and advance the child's quality of life. Pediatric Nursing Excellence (PNE) model assist nurses in providing the optimal care possible to children, their work environments, also to recognize their efforts to enhance childcare through system improvement. Also, the nursing excellence model provide nurses the necessary knowledge and practice to deliver high-quality nursing care. as well to carry out their responsibilities efficiently and to identify the recent trends in specialty nursing excellence.

The present study aims to evaluate application of pediatric nursing excellence model on nurses' performance regarding care of children undergoing orthopedic surgeries

Hypotheses:

Nurses that participate in the pediatric nursing excellence model application are expected to increase their performance when caring for children having orthopedic surgery.

Design A randomized controlled trial with two parallel groups Randomization Participants will be randomly assigned to either the intervention or control group (50 per group) using a computer-generated randomization sequence with block sizes of varying lengths to ensure allocation concealment.

The study will be conducted in the pediatric inpatient surgical unit at Tanta University Hospital which is affiliated to the ministry of higher education and scientific research.

Three tools will be employed to obtain the relevant data to the present study. Tool (I): Nurses, knowledge assessment questionnaire Part (1): Nurses, Socio demographic characteristics: such as age, gender, academic qualifications, years of experience at the surgical unit, and previous training courses regarding care of children undergoing orthopedic surgeries.

Part (2): Nurses, knowledge Assessment This part assessed nurses, knowledge regarding orthopedic surgeries which included types, causes, complications and diagnostic methods.

Part (3) Nurses knowledge regarding preoperative and post operative nursing care. It included preoperative care as (assess general body condition, vital signs, intake and output, measurement of weight, investigations and diagnostic tests), postoperative nursing care as: complications after surgery, precautions to prevent infection, pain management, wound care, intake and output, discharge instructions.

Scoring system: Each item was scored as follows: correct answers scored (2), correct and incomplete scored (1) and the incorrect or do not know answers scored (0).

The nurses' total knowledge was classified as the following:

* ≥ 80% was considered high level of knowledge
* 60-80 was considered moderate level of knowledge
* <60 was considered low level of knowledge Tool (II): Orthopedic surgeries Nurses, practice observational checklist Part I: Nursing care for children on admission: hand washing procedure, vital signs, weight measurement, laboratory sampling, care of intravenous infusion.

Part II: Preoperative nursing care which includes psychological preparation, parent and child education, informed consent, physical preparation and safety precautions.

Part III: post-operative nursing care; immediately post-operative nursing care, Discharge from the recovery room, pain management, post-operative first day nursing care, wound care, discharge instructions for parents and child.

Scoring system: Each step was evaluated as follows.

* Done correctly scored (1 point)
* Not done scored zero
* Total practice scores are transformed into percentages.
* ≥ 80% considered satisfactory practice.
* <80% considered unsatisfactory practice. Tool III: Pediatric nursing excellence (PNE) model, adopted from McDowell et al., (2023). It will be written in an Arabic language and consisted of (15) Likert-type questions to assess nurses' general excellence level regarding the care of children undergoing orthopedic surgeries grouped under five main categories including engagement, values, principles, care delivery and continuous improvement. Each one of these categories had 3 sub items as following: Engagement: [collaboration, professionalism, and professional development], Values [advocacy, ethics, and quality of life], Principles [equity, holistic care and family centered care], Care delivery [care coordination, care planning and health promotion] and Continuous improvement [evidence-based practice, outcomes, and quality standards]. Scoring system for nurses' excellence level: The nurses excellence level was evaluated from 0 to 30 as; low excellence level 0-9, moderate excellence level 10-19, high excellence level 20-30. The questionnaire rating through a 3-point Likert scale, including agree (2), neutral (1), and disagree (0).

Data collection procedure: through three phases:

I-Assessment Phase:

It will be carried out by the researchers for all nurses to assess nurses, sociodemographic characteristics and knowledge about Tool I

* Nurses practice regarding oral care of mechanically ventilated children will be assessed before, immediate and after one month of program implementation using Tool II
* Nurses will be interviewed individually or in group to fill the questionnaire sheet.

II-Implementation Phase:

-The educational intervention will be prepared and conducted in the previously mentioned settings during the morning shift through four sessions.

The sessions will cover the following topics

* The first session: types, causes, complications and diagnostic methods
* The second session: preoperative and post operative nursing care for children undergoing orthopedic surgeries
* The third session: Pediatric excellence model and its intended purposes, components, general application,
* The fourth session: Excellence criteria of nursing care for child safety, and prevention of medication errors. Approaches for promoting nursing excellence identification in the practice area.
* The quality requirements in managing human and material resources including equipment handling and nursing care. Latest trends in health care services affecting nursing care provided for children undergoing orthopedic surgeries

III-Evaluation phase:

Evaluation of pediatric nursing excellence model on nurses, performance regarding care of children undergoing orthopedic surgeries will be done through comparing the pre and posttest. This phase will be done three times before, immediately and one month later.

ELIGIBILITY:
Inclusion Criteria:

* Nurses with a Diploma or bachelor's degree or higher
* No present or previous participation in the same study
* Willing to give written informed consent to participate in the study.

Exclusion Criteria:

* present or previous participation in the same study
* Not Willing to give written informed consent to participate in the study.
* Missing two sessions

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Nurses performance | six months study period
  High Level of Knowledge: ≥ 80 % • Using Nurses, knowledge Assessment that will assess nurses, knowledge regarding orthopedic surgeries which included types, causes, complications and diagnostic methods as well as Nurses' knowledge regarding preoperative and post operative nursing care.
  Satisfactory level practice: ≥ 80%
  * Using practice observational checklist that includes Nursing care for children on admission: hand washing procedure, vital signs, weight measurement, laboratory sampling, care of intravenous infusion. Preoperative nursing care which includes psychological preparation, parent and child education, informed consent, physical preparation and safety precautions
  High Level of excellence: ≥ 75 %
  • Using Pediatrics Nursing Excellence Model (PNE)- model that include collaboration, professionalism, advocacy, ethics, Principles of equity, holistic care and family centered care.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Department of New Surgical Hospital, and Pediatric Surgical Orthopedic Department - Tanta University Hospital., Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
1. No personal identification data will be collected, so the researchers assure participants anonymity.
  2. The researchers will collect only the data required to this study.
  3. Demographic data of participants will be coded to maintain confidentiality.
  4. All submitted data are saved and handled electronically by the researchers only through password-protected files.